CLINICAL TRIAL: NCT00369629
Title: Phase I/II Trial of Gemcitabine/Pemetrexed Combination in Patients With Advanced Cutaneous T-Cell Lymphoma
Brief Title: Gemcitabine and Pemetrexed Disodium in Treating Patients With Advanced Mycosis Fungoides or Sézary Syndrome
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This was planned as a phase I/II study originally, but due to a lack of funding, the phase II portion was never conducted.
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 05H8; P30CA060553 (NIH); STU00006771 (Other: Northwestern University IRB)
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Lymphoma
Keywords: recurrent mycosis fungoides/Sezary syndrome; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Mycosis Fungoides; Sezary Syndrome; Lymphoma, T-Cell, Cutaneous | interventions — Gemcitabine; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 (Experimental): Pemetrexed at a dose of 400 mg/m2 will be given to patients on day 1 and day 15 of 28 day cycle.
  Gemcitabine at a dose of 800 mg/m2 will be given following pemetrexed on day 1 and 15 of a 28-day cycle.
  Interventions: Drug: Gemcitabine; Drug: Pemetrexed
- Cohort 2 (Experimental): Pemetrexed at a dose of 500 mg/m2 will be given to patients on day 1 and day 15 of 28 day cycle.
  Gemcitabine at a dose of 800 mg/m2 will be given following pemetrexed on day 1 and 15 of a 28-day cycle.
  Interventions: Drug: Gemcitabine; Drug: Pemetrexed
- Cohort 3 (Experimental): Pemetrexed at a dose of 500 mg/m2 will be given to patients on day 1 and day 15 of 28 day cycle.
  Gemcitabine at a dose of 1000 mg/m2 will be given following pemetrexed on day 1 and 15 of a 28-day cycle.
  Interventions: Drug: Gemcitabine; Drug: Pemetrexed
- Cohort 4 (Experimental): Pemetrexed at a dose of 500 mg/m2 will be given to patients on day 1 and day 15 of 28 day cycle.
  Gemcitabine at a dose of 1200 mg/m2 will be given following pemetrexed on day 1 and 15 of a 28-day cycle.
  Interventions: Drug: Gemcitabine; Drug: Pemetrexed

INTERVENTIONS:
Drug: Gemcitabine — Patients will be treated in cohorts of 3-6 per cohort. The starting dose of gemcitabine will be 800 mg/m^2 given as an intravenous (IV) infusion on days 1 and 15 of each 28-day cycle. The dose will be escalated for each subsequent cohort of patients, up to a maximum of 1200 mg/m^2.
Drug: Pemetrexed — Patients will be treated in cohorts of 3-6 per cohort. The starting dose of pemetrexed will be 400 mg/m^2 given as an intravenous (IV) infusion on days 1 and 15 of each 28-day cycle. The dose will be escalated for each subsequent cohort of patients, up to a maximum of 500 mg/m^2.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Pemetrexed disodium may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving gemcitabine together with pemetrexed disodium may kill more cancer cells.

PURPOSE: This was planned as a phase I/II trial studying the side effects and determining the best dose of gemcitabine hydrochloride when given together with pemetrexed disodium. Unfortunately, due to a lack of funding, the phase II portion was never conducted.

DETAILED DESCRIPTION:
OBJECTIVES:

1. Determine the safety and tolerability of gemcitabine hydrochloride and pemetrexed disodium in patients with advanced mycosis fungoides or Sézary syndrome. (Phase I)
2. Determine the maximum tolerated dose of gemcitabine hydrochloride when administered with pemetrexed disodium in these patients. (Phase I)

OUTLINE: This is a phase I, dose-escalation study of gemcitabine hydrochloride. Originally, this was designed to be followed by a phase II portion to determine the efficacy in this population. Unfortunately, due to a lack of funding, the phase II portion was never conducted.

During Phase I: Patients receive pemetrexed disodium IV over 10 minutes and gemcitabine hydrochloride IV on days 1 and 15. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of gemcitabine hydrochloride until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which ≥ 2 of 6 patients experience dose-limiting toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed* mycosis fungoides or Sézary syndrome

  * Stage IB-IVB disease NOTE: *Pathology report must read diagnostic or consistent with mycosis fungoides/Sézary syndrome
* Failed ≥ 1 prior systemic treatment
* Measurable disease

  * At least 1 indicator lesion must be designated prior to study entry

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 6 months
* Creatinine ≤ 2.0 mg/dL
* Creatinine clearance ≥ 45 mL/min
* Bilirubin ≤ 2.2 mg/dL
* AST and ALT ≤ 2 times upper limit of normal
* WBC ≥ 3,000/mm³
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* No acute infection requiring systemic treatment
* No history of severe hypersensitivity reaction to the study drugs or to any other ingredient used in their formulation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 4 weeks since prior topical therapy, systemic chemotherapy, or biological therapy
* No acetylsalicylic acid or other nonsteroidal anti-inflammatory drugs (NSAIDs) for 2 days before and for 2 days after pemetrexed disodium infusion (5 days before and for 2 days after pemetrexed disodium infusion for patients taking NSAIDs with a long half-life [e.g., naproxen, refocoxib, or celecoxib])
* No concurrent topical agents except emollients
* No other concurrent topical or systemic anticancer therapies
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-08-28 (Actual); Primary Completion 2012-07-16 (Actual); Study Completion 2013-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Pro, MD, Principal Investigator — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened for accrual on June 6, 2006 in phase I with a 3+3 cohort design to find the recommended phase II dose. Phase II would expand to enroll a total of 20 evaluable patients at the recommended dose. The study was closed permanently on September 12, 2012 after 14 patients had been enrolled in the phase I part.
Groups:
- Cohort 1: Patients will be treated in cohorts of 3-6 per cohort in a dose escalation of pemetrexed and gemcitabine
  Pemetrexed at a dose of 400 mg/m2 will be given to patients on day 1 and day 15 of 28 day cycle.
  Gemcitabine at a dose of 800 mg/m2 will be given following pemetrexed on day 1 and 15 of a 28-day cycle.
- Cohort 2: Patients will be treated in cohorts of 3-6 per cohort in a dose escalation of pemetrexed and gemcitabine
  Pemetrexed at a dose of 500 mg/m2 will be given to patients on day 1 and day 15 of 28 day cycle.
  Gemcitabine at a dose of 800 mg/m2 will be given following pemetrexed on day 1 and 15 of a 28-day cycle.
- Cohort 3: Patients will be treated in cohorts of 3-6 per cohort in a dose escalation of pemetrexed and gemcitabine
  Pemetrexed at a dose of 500 mg/m2 will be given to patients on day 1 and day 15 of 28 day cycle.
  Gemcitabine at a dose of 1000 mg/m2 will be given following pemetrexed on day 1 and 15 of a 28-day cycle.
- Cohort 4: Patients will be treated in cohorts of 3-6 per cohort in a dose escalation of pemetrexed and gemcitabine
  Pemetrexed at a dose of 500 mg/m2 will be given to patients on day 1 and day 15 of 28 day cycle.
  Gemcitabine at a dose of 1200 mg/m2 will be given following pemetrexed on day 1 and 15 of a 28-day cycle.
Period: Treated 2 Cycles/Reached First Response
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 6 | 3 | 5 | 0 (No patients were enrolled at this dose level as the study closed early due to lack of funding.)
Completed | 4 | 2 | 3 | 0
Not Completed | 2 | 1 | 2 | 0
Not completed — Physician Decision | 0 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Progressive disease | 2 | 0 | 0 | 0
Period: Moved on to 4 More Cycles
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 4 | 2 | 3 | 0
Completed | 4 | 2 | 2 | 0
Not Completed | 0 | 0 | 1 | 0
Not completed — Progressive Disease | 0 | 0 | 1 | 0
Period: Completed 4 More Cycles
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 4 | 2 | 2 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 4 | 2 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 0
Not completed — Progressive disease | 2 | 1 | 2 | 0
Period: Follow up for 1 Year
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 6 (All patients treated on study go into the follow up period) | 3 | 5 | 0
Completed | 4 | 1 | 2 | 0
Not Completed | 2 | 2 | 3 | 0
Not completed — Death | 2 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — stopped being followed as study closed | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Gemcitabine and Pemetrexed Disodium: Gemcitabine: Patients will be treated in cohorts of 3-6 per cohort. The starting dose of gemcitabine will be 800 mg/m^2 given as an intravenous (IV) infusion on days 1 and 15 of each 28-day cycle. The dose will be escalated for each subsequent cohort of patients, up to a maximum of 1200 mg/m^2.
  Pemetrexed: Patients will be treated in cohorts of 3-6 per cohort. The starting dose of pemetrexed will be 400 mg/m^2 given as an intravenous (IV) infusion on days 1 and 15 of each 28-day cycle. The dose will be escalated for each subsequent cohort of patients, up to a maximum of 500 mg/m^2.
Arm/Group | Gemcitabine and Pemetrexed Disodium
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose as Measured by the Number of Dose Limiting Toxicities Seen in Cohort.
Description: Only dose limiting toxicities (DLT) were collected. DLTs were graded according to the National Cancer Institute's Common Toxicity Criteria for adverse events version 3.0 (CTCAE v3.0) according to the following:
  Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE
  The occurrence of any of the following toxicities during the first treatment cycle constitutes DLT in this study:
  Grade 3 and/or 4 non-hematologic toxicity other than grade 3 nausea or vomiting.
  Grade 3 and/or 4 unexpected non-hematologic toxicities. Grade 4 vomiting despite maximal antiemetic support. Grade 4 neutropenia and fever during first cycle. Grade 4 neutropenia on Day 1 of 2nd treatment cycle despite growth factor support or grade 4 thrombocytopenia on Day 1 of 2nd treatment cycle.
Time Frame: From the day that the first treatment is given through the first 28 day period for each patient.
Population: Patients that experienced a DLT in the first cycle in each cohort. If one DLT is seen in the first 3 patients then 3 more patients are enrolled in that cohort. MTD and is defined as the lowest dose level at which two or more patients experience a DLT. The study closed before enough patients were enrolled to determine the MTD or define DLTs.
Measure: Number; unit: DLT
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 6 | 3 | 5 | 0
DLT
  Perforated sigmoid diverticulitis | 1 | 0 | 0 |
  Febrile neutropenia | 0 | 0 | 1 |

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a 6 year period for the study. Adverse events were collected from the start of treatment every 14 days until 30 days after the last treatment, for a maximum of 6 cycles. 1 cycle =28 days.
Description: Adverse events were collected every 14 days on a 28 day cycle from the start of treatment until 30 days after the last dose for a maximum of 6 cycles of treatment.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
All-Cause Mortality (participants affected / at risk) | 5/6 | 2/3 | 2/5 | 0/0
Serious Adverse Events (participants affected / at risk) | 2/5 | 0/3 | 1/5 | 0/0
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 5/5 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=5) | Cohort 2 (N=3) | Cohort 3 (N=5) | Cohort 4 (N=0)
Perforated sigmoid diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteremia CMV (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Line sepsis and neutropenia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=6) | Cohort 2 (N=3) | Cohort 3 (N=5) | Cohort 4 (N=0)
allergic rhinitis (Immune system disorders) | 0 | 1 | 0 | 0
Otitis, external ear (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Hemoglobin (Blood and lymphatic system disorders) | 6 | 2 | 4 | 0
Neutrophils (neutropenia) (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Leukocytes (total white blood cells) (Blood and lymphatic system disorders) | 3 | 1 | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 5 | 1 | 4 | 0
Platelets (thrombocytopenia) (Blood and lymphatic system disorders) | 4 | 1 | 2 | 0
Hypotension (Cardiac disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 1 | 0
Fatigue (General disorders) | 2 | 3 | 4 | 0
Fever (General disorders) | 1 | 0 | 3 | 0
Insomnia (General disorders) | 0 | 1 | 0 | 0
Rigor/chills (General disorders) | 0 | 0 | 1 | 0
Sweating/diaphoresis (General disorders) | 0 | 0 | 1 | 0
Weight loss (General disorders) | 0 | 1 | 0 | 0
International normalized Ration of prothrombin time (INR) (Investigations) | 0 | 0 | 1 | 0
Flushing (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Hair loss (alopecia) (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Pruritus/itching (Skin and subcutaneous tissue disorders) | 4 | 1 | 1 | 0
Anorexia (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 4 | 0
Dehydration (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 3 | 0
Heartburn/dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 2 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 3 | 0
Hemorrhage, GU: Urinary NOS (Renal and urinary disorders) | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0
Dermatitis (Infections and infestations) | 1 | 0 | 0 | 0
Colitis, infectious (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
MRSA (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Edema, Limb (Blood and lymphatic system disorders) | 1 | 0 | 4 | 0
Edema (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Edema, trunk/genital (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Alkaline phosphatase (Metabolism and nutrition disorders) | 4 | 0 | 0 | 0
ALT increase (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0
AST increase (Metabolism and nutrition disorders) | 4 | 2 | 3 | 0
Albumin, serum-low (Metabolism and nutrition disorders) | 4 | 1 | 5 | 0
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Creatinine (Metabolism and nutrition disorders) | 5 | 1 | 2 | 0
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 4 | 3 | 4 | 0
Glucose, Serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Sodium, serum low (hyponatremia) (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0
Sensory Neuropathy (Nervous system disorders) | 0 | 0 | 2 | 0
Mental status (Nervous system disorders) | 1 | 0 | 1 | 0
Anxiety (mood alteration) (Nervous system disorders) | 0 | 1 | 0 | 0
Depression (mood alteration) (Nervous system disorders) | 0 | 1 | 0 | 0
Abdomen pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Limb pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Scrotum pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Urethra pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Pain NOS (General disorders) | 0 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Shortness of breath (dyspnea) (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Blurred vision (Eye disorders) | 1 | 0 | 0 | 0
Watery eye (epiphora, tearing) (Eye disorders) | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was terminated early before the last patient was enrolled in phase I due to lack of funding. The phase II portion was never conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes